CLINICAL TRIAL: NCT02563067
Title: A 52-week, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of QAW039 When Added to Existing Asthma Therapy in Patients With Uncontrolled Severe Asthma.
Brief Title: Study of Efficacy and Safety of QAW039 in Patients With Severe Asthma Inadequately Controlled With Standard of Care Asthma Treatment.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAW039A2314; 2015-003172-67 (EudraCT Number)
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Results first posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Asthma
Keywords: Asthma; QAW039
MeSH Terms: conditions — Asthma | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- QAW039 150 mg (Experimental): QAW039 150 mg once daily
  Interventions: Drug: QAW039
- QAW039 450 mg (Experimental): QAW039 450 mg once daily
  Interventions: Drug: QAW039
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: QAW039 — QAW039 150 mg once daily
  Arms: QAW039 150 mg
Drug: QAW039 — QAW039 450 mg once daily
  Arms: QAW039 450 mg
Drug: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
This study aimed to determine the efficacy and safety of QAW039 and QAW039 450 mg compared to placebo, when added to GINA (Global Initiative for Asthma) steps 4 and 5 standard-of- care (SoC) asthma therapy (GINA 2016) in the following two populations:

* patient with inadequately controlled severe asthma and high eosinophil counts (eosinophil count at Visit 1 ≥250 cells/ µl) (sub-population)
* patients with inadequately controlled severe asthma (overall study population) Inadequate control is defined as partly controlled or uncontrolled asthma (GINA 2016)

DETAILED DESCRIPTION:
This study used a randomized, multicenter, double-blind, placebo-controlled parallel-group design in which QAW039 (150 mg and 450 mg) or placebo was added to GINA steps 4 and 5 asthma therapy.

The study included:

* Screening period of up to 2 weeks to assess eligibility;
* Run-in period of approximately 2 weeks and a maximum of 6 weeks on placebo to collect baseline data for efficacy variables and compliance with the Electronic Peak Flow/ eDiary device. Upon completion of the run-in period, all patients who met the eligibility criteria were randomized to one of three treatments: QAW039 150 mg or QAW039 450 mg or placebo once daily in a ratio of 1:1:1.
* Treatment period of 52 weeks (assessment period for all Primary and Secondary Outcome Measures). Clinic visits were scheduled approximately 4 weeks after randomization and then at approximately 8-week intervals during the active-treatment period. Phone calls occurred at specified time points between visits occurring at 8-week intervals. Patients who had successfully completed 52 weeks of treatment in this study were offered an optional participation in a safety study (CQAW039A2315).
* Follow-up period of 4 weeks, investigational and drug-free, following the last dose of study drug. A follow-up visit occurred approximately 4 weeks (i.e., approximately 30 days) following the last dose of study therapy to complete safety assessments and pregnancy testing (if applicable).

The follow-up period applied to all patients except those patients who had entered the optional safety study (CQAW039A2315) directly after the Week 52 study visit

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male and female patients aged ≥12 years.
* A diagnosis of severe asthma, uncontrolled on GINA 4/5 asthma medication.
* Evidence of airway reversibility or airway hyper- reactivity.
* FEV1 ≤80% of the predicted normal value for patients aged ≥18 years; FEV1 of ≤90% for patients aged 12 to <18 years
* An ACQ score ≥1.5
* A history of 2 or more asthma exacerbations within the 12 months prior to entering the study.

Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives of study entry, or within 30 days, whichever is longer.
* Subjects who have participated in another trial of QAW039.
* A QTcF (Fridericia) ≥450 msec (male) or ≥460 msec (female).
* History of malignancy with the exception of local basal cell carcinoma of the skin.
* Pregnant or nursing (lactating) women.
* Serious co-morbidities.
* Patients on >20 mg of simvastatin, > 40 mg of atorvastatin, >40 mg of pravastatin, or >2 mg of pitavastatin.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 877 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (144):
- United States (17):
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Winter Park, Florida
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Edmond, Oklahoma
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, Richmond, Virginia
- Argentina (13):
  - Novartis Investigative Site, Berazategui, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Ranelagh, Partido de Berazate, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, Santa Rosa, La Pampa Province
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Santa Fe
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Vancouver BC, British Columbia
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec
- Czechia (7):
  - Novartis Investigative Site, Jindřichův Hradec, Czech Republic
  - Novartis Investigative Site, Teplice, Czech Republic
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Karlovy Vary
  - Novartis Investigative Site, Mladá Boleslav
  - Novartis Investigative Site, Plzen-Bory
- Greece (3):
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- India (9):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
- Italy (20):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Acquaviva delle Fonti, BA
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Cagliari, Sicily
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Legnago, VR
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Reggio Emilia
  - Novartis Investigative Site, Salerno
- Japan (16):
  - Novartis Investigative Site, Chikushino-shi, Fukuoka
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Naka-gun, Ibaraki
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Hamamatsu, Shizuoka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Setagaya-Ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima Ku, Tokyo
- Lebanon (3):
  - Novartis Investigative Site, El Chouf, LBN
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
- Malaysia (4):
  - Novartis Investigative Site, Kota Bharu, Kelantan
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, Taiping, Perak
  - Novartis Investigative Site, Batu Caves
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Guadalajara Jalisco, Jalisco
  - Novartis Investigative Site, Zapopan, Jalisco
- Netherlands (4):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Leiden
- Russia (8):
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Stavropol
  - Novartis Investigative Site, Yekaterinburg
- Serbia (2):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Kragujevac
- Slovakia (10):
  - Novartis Investigative Site, Dúbravka, Bratislava Region
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Liptovský Hrádok, Slovak Republic
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Spišská Nová Ves
  - Novartis Investigative Site, Vyšné Hágy
- South Africa (3):
  - Novartis Investigative Site, Tygerberg, Cape Town
  - Novartis Investigative Site, Mowbray
  - Novartis Investigative Site, Panorama
- Spain (12):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Jerez de la Frontera, Cadiz
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sabadell, Catalonia
  - Novartis Investigative Site, Lugo, Galicia
  - Novartis Investigative Site, Girona
  - Novartis Investigative Site, Guadalajara
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Santiago de Compostela
  - Novartis Investigative Site, Zaragoza
- Taiwan (2):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Taichung

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Brightling CE, Gaga M, Inoue H, Li J, Maspero J, Wenzel S, Maitra S, Lawrence D, Brockhaus F, Lehmann T, Brindicci C, Knorr B, Bleecker ER. Effectiveness of fevipiprant in reducing exacerbations in patients with severe asthma (LUSTER-1 and LUSTER-2): two phase 3 randomised controlled trials. Lancet Respir Med. 2021 Jan;9(1):43-56. doi: 10.1016/S2213-2600(20)30412-4. Epub 2020 Sep 24. PMID 32979986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from centers in Argentina (18), Canada (5), Czech Republic (7), Greece (6), India (12), Israel (5), Italy (22), Japan (16), Lebanon (3), Malaysia (4), Mexico (3), Netherlands (4), Russian Federation (11), Serbia (4), Slovakia (11), South Africa (3), Spain (13), Taiwan (3) and the United States (19).
Pre-assignment Details: The study included a Screening period of up to 2 weeks and a Placebo Run-in period of 2 to 6 weeks, during which eligibility for randomization was determined
Period: Overall Study
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Started | 296 | 294 | 287
FAS/SAF: High Eosinophils Subpopulation (Full analysis set/safety set. All patients who received study drug and had high eosinophils count) | 198 | 196 | 193
FAS/SAF: Overall Population (Full analysis set/safety set. All patients who received study drug) | 296 | 293 | 287
Completed | 277 | 268 | 267
Not Completed | 19 | 26 | 20
Not completed — Subject/guardian decision | 14 | 20 | 16
Not completed — Physician Decision | 0 | 1 | 3
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Technical problems | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Death | 0 | 1 | 1
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Death post Treatment/safety period | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo | Total
Number analyzed (Participants) | 296 | 294 | 287 | 877
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (14.60) | 49.6 (15.25) | 50.9 (14.16) | 50.1 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 165 | 178 | 177 | 520
  Male | 131 | 116 | 110 | 357
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 234 | 235 | 227 | 696
  Black | 6 | 4 | 1 | 11
  Asian | 44 | 41 | 41 | 126
  Native American | 2 | 2 | 4 | 8
  Unknown | 2 | 2 | 3 | 7
  Other | 8 | 10 | 11 | 29

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate-to-severe Asthma Exacerbations During the 52-week Treatment Period in High Eosinophils Subpopulation
Description: A severe asthma exacerbation is defined as treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days and hospitalization; or treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days and emergency department visit (greater than 24 hours*); or death due to asthma.
  A moderate asthma exacerbation is defined as treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days either as an outpatient or in emergency department visits (Emergency department visit less than or equal to 24 hours). The high eosinophils subpopulation consists of all patients with blood eosinophil count ≥ 250 cells/μL at baseline.
Time Frame: 52 weeks
Population: Full Analysis Set (FAS) in high eosinophils subpopulation (count ≥ 250 cells/μL)
Measure: Least Squares Mean (95% Confidence Interval); unit: Events/year
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 198 | 196 | 193
Events/year | 0.73 [0.57 to 0.94] | 0.76 [0.59 to 0.99] | 1.06 [0.84 to 1.33]
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.059, negative binomial regression model; adjusted p-value, closed testing procedure across the primary and key secondary null hypotheses. Overall type I error rate controlled at two-sided 5%; Rate Ratio = 0.69, 95% CI 2-sided [0.50 to 0.96]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.114, negative binomial regression model; [statistical method as in outcome 1, analysis 1]; Rate Ratio = 0.72, 95% CI 2-sided [0.52 to 1.01]

2. Secondary Outcome: Change From Baseline to Week 52 in Asthma Quality of Life Questionnaire for Participants 12 Years and Older (AQLQ+12) Score in High Eosinophils Subpopulation
Description: AQLQ is a 32-item instrument administered as a self-assessment. AQLQ+12 is a modified version of AQLQ developed to measure functional impairments of participants aged 12-70 years. It is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Participants were asked to recall their experiences during the last 2 weeks and respond to each question on a 7-point scale (1=severe impairment, 7=no impairment), where higher scores indicated "better quality of life." Overall AQLQ+12 score is the mean of all 32 responses. The high eosinophils subpopulation consists of all patients with blood eosinophil count ≥ 250 cells/μL at baseline.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) in high eosinophils subpopulation (count ≥ 250 cells/μL)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 198 | 196 | 193
units on a scale | 0.73 (0.061) | 0.71 (0.062) | 0.58 (0.062)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.369, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.02 to 0.32]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.824, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.13, 95% CI 2-sided [-0.04 to 0.30]

3. Secondary Outcome: Change From Baseline to Week 52 in Asthma Control Questionnaire-5 (ACQ-5) Score in High Eosinophils Subpopulation
Description: The ACQ-5 is a five-item, self-completed questionnaire, which is used as a measure of asthma control of a participant. The five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) enquire about the frequency and/or severity of symptoms over the previous week. The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/ limitation) scale. The ACQ-5 score is the average of the individual item scores and ranges from 0 to 6. Higher scores indicates worsening of condition. The high eosinophils subpopulation consists of all patients with blood eosinophil count ≥ 250 cells/μL at baseline.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) in high eosinophils subpopulation (count ≥ 250 cells/μL)
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 198 | 196 | 193
units on a scale | -0.92 (0.067) | -0.84 (0.068) | -0.75 (0.069)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.369, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.36 to 0.01]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.824, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.28 to 0.10]

4. Secondary Outcome: Change From Baseline to Week 52 in Pre-dose Forced Expiratory Volume in 1 Second (FEV1) in High Eosinophils Subpopulation
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline is defined as the last available FEV1 measurement taken prior to the first dose of randomized study drug. The high eosinophils subpopulation consists of all patients with blood eosinophil count ≥ 250 cells/μL at baseline.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS) in high eosinophils subpopulation (count ≥ 250 cells/μL)
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 198 | 196 | 193
Liter | 0.192 (0.0306) | 0.162 (0.0311) | 0.124 (0.0313)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.369, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.068, 95% CI 2-sided [-0.018 to 0.154]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.824, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.038, 95% CI 2-sided [-0.048 to 0.124]

5. Primary Outcome: Rate of Moderate-to-severe Asthma Exacerbations During the 52-week Treatment Period in Overall Population
Description: A severe asthma exacerbation is defined as treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days and hospitalization; or treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days and emergency department visit (greater than 24 hours*); or death due to asthma.
  A moderate asthma exacerbation is defined as treatment with 'rescue' systemic corticosteroids for greater than or equal to 3 days either as an outpatient or in emergency department visits (Emergency department visit less than or equal to 24 hours).
Time Frame: 52 weeks
Population: Full Analysis Set (FAS), including all randomized patients who received at least one dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Events/year
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 296 | 293 | 287
Events/year | 0.76 [0.62 to 0.92] | 0.70 [0.57 to 0.87] | 0.93 [0.76 to 1.12]
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.369, negative binomial regression model; [statistical method as in outcome 1, analysis 1]; Rate Ratio = 0.82, 95% CI 2-sided [0.62 to 1.07]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.348, negative binomial regression model; [statistical method as in outcome 1, analysis 1]; Rate Ratio = 0.76, 95% CI 2-sided [0.58 to 1.00]

6. Secondary Outcome: Change From Baseline to Week 52 in Asthma Quality of Life Questionnaire for Participants 12 Years and Older (AQLQ+12) Score in Overall Population
Description: AQLQ is a 32-item instrument administered as a self-assessment. AQLQ+12 is a modified version of AQLQ developed to measure functional impairments of participants aged 12-70 years. It is divided into 4 domains: activity limitation, symptoms, emotional function, and environmental stimuli. Participants were asked to recall their experiences during the last 2 weeks and respond to each question on a 7-point scale (1=severe impairment, 7=no impairment), where higher scores indicated "better quality of life." Overall AQLQ+12 score is the mean of all 32 responses.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS), including all randomized patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 296 | 293 | 287
units on a scale | 0.62 (0.050) | 0.67 (0.050) | 0.55 (0.051)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.824, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.07 to 0.21]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.824, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.02 to 0.26]

7. Secondary Outcome: Change From Baseline to Week 52 in Asthma Control Questionnaire-5 (ACQ-5) Score in Overall Population
Description: The ACQ-5 is a five-item, self-completed questionnaire, which is used as a measure of asthma control of a participant. The five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) enquire about the frequency and/or severity of symptoms over the previous week. The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/ limitation) scale. The ACQ-5 score is the average of the individual item scores and ranges from 0 to 6. Higher scores indicates worsening of condition.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS), including all randomized patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 296 | 293 | 287
units on a scale | -0.83 (0.055) | -0.77 (0.055) | -0.70 (0.055)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.824, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.28 to 0.03]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.824, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.23 to 0.08]

8. Secondary Outcome: Change From Baseline to Week 52 in Pre-dose Forced Expiratory Volume in 1 Second (FEV1) in Overall Population
Description: Forced Expiratory Volume in one second (FEV1) is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Baseline is defined as the last available FEV1 measurement taken prior to the first dose of randomized study drug.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS), including all randomized patients who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 296 | 293 | 287
Liter | 0.153 (0.0247) | 0.164 (0.0249) | 0.103 (0.0250)
Statistical Analysis 1: Comparison: QAW039 150 mg vs Placebo; Test type: Superiority; p = 0.369, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.050, 95% CI 2-sided [-0.019 to 0.119]
Statistical Analysis 2: Comparison: QAW039 450 mg vs Placebo; Test type: Superiority; p = 0.595, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.061, 95% CI 2-sided [-0.008 to 0.130]

9. Post Hoc Outcome: All Collected Deaths
Description: Total Deaths are presented from first dose of study treatment until discontinuation of trial, up to maximum duration of 56 weeks.
  Deaths on-treatment are presented from first dose of study treatment until last dose of study treatment plus 30 days, up to maximum duration of 56 weeks.
Time Frame: up to 56 weeks
Population: Safety Set (SAF), including all randomized patients who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
Number analyzed (Participants) | 296 | 293 | 287
Participants
  Total Deaths | 1 | 1 | 1
  Deaths on-treatment | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are presented from first dose of study treatment until last dose of study treatment plus 7 days post treatment. Serious AEs (including the All-Cause Mortality data table) are presented from first dose of study treatment until last dose of study treatment plus 30 days post treatment, up to maximum duration of 56 weeks.
Description: Any sign or symptom that occurs during the study treatment plus 7 days post treatment for adverse events and 30 days post treatment for serious adverse events.
Groups:
- QAW039 150 mg: QAW039 150 mg
- QAW039 450 mg: QAW039 450 mg
- Placebo: Placebo
Arm/Group | QAW039 150 mg | QAW039 450 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/296 | 1/293 | 1/287
Serious Adverse Events (participants affected / at risk) | 20/296 | 20/293 | 18/287
Other Adverse Events (participants affected / at risk) | 181/296 | 183/293 | 180/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=296) | QAW039 450 mg (N=293) | Placebo (N=287)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 4 | 3
Sinusitis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain hypoxia (Nervous system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Uterine enlargement (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QAW039 150 mg (N=296) | QAW039 450 mg (N=293) | Placebo (N=287)
Bronchitis (Infections and infestations) | 37 | 30 | 32
Influenza (Infections and infestations) | 17 | 18 | 13
Nasopharyngitis (Infections and infestations) | 33 | 42 | 26
Rhinitis (Infections and infestations) | 10 | 15 | 13
Upper respiratory tract infection (Infections and infestations) | 18 | 16 | 14
Upper respiratory tract infection bacterial (Infections and infestations) | 10 | 8 | 14
Viral upper respiratory tract infection (Infections and infestations) | 20 | 28 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 5 | 9
Headache (Nervous system disorders) | 19 | 21 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 129 | 119 | 145
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT02563067/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02563067/SAP_001.pdf